CLINICAL TRIAL: NCT02947867
Title: Prospective, Randomised, Placebo-controlled, Double-masked, Three-armed Multi-centre Trial of Aganirsen Versus Vehicle in Patients After Ischaemic Central Retinal Vein Occlusion With a High Risk to Develop Neovascular Glaucoma
Brief Title: Trial of Aganirsen in iCRVO Patients at Risk of Developing NVG
Acronym: STRONG
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gene Signal SAS (Industry)
Collaborators: Johannes Gutenberg University Mainz (Other); University Hospital of Cologne (Other); Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-101-P1-NVR; 2014-000239-18 (EudraCT Number)
Record Dates: First submitted 2016-10-15; First posted 2016-10-28 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Ischaemic Central Retinal Vein Occlusion; Neovascular Glaucoma
MeSH Terms: conditions — Glaucoma, Neovascular | interventions — GS 101

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- aganirsen "low-dose": (Experimental): 43µg daily, one drop of 0.86 mg/g emulsion (morning) + one drop of placebo (evening) daily
  Interventions: Drug: aganirsen
- aganirsen "high-dose" (Experimental): 86µg daily, one drop of 0.86 mg/g emulsion twice daily (morning and evening)
  Interventions: Drug: aganirsen
- aganirsen placebo (vehicle) (Placebo Comparator): one drop of placebo emulsion (morning) + one drop of placebo emulsion (evening) daily
  Interventions: Drug: aganirsen

INTERVENTIONS:
Drug: aganirsen — aganirsen antisense oligonucleotide against Insulin Receptor Substrate (IRS-1)
  Other Names: GS-101

SUMMARY:
A prospective, randomised, placebo-controlled, double-masked, three-armed multi-centre phase II/III trial for the Study of a Topical Treatment of Ischaemic Central Retinal Vein Occlusion to Prevent Neovascular Glaucoma - the STRONG Study

DETAILED DESCRIPTION:
The STRONG Study is a phase II/III prospective, randomised, placebo-controlled, double-masked, three-armed multi-centre study of aganirsen antisense oligonucleotide, a topical treatment for iCRVO intended to prevent Neovascular Glaucoma (NVG). The study will evaluate the efficacy of two different doses of aganirsen formulated in an eye emulsion in avoiding new vessel formation by blocking the Insulin Receptor Substrate (IRS)-1. Eligible patients will be treated with aganirsen or placebo for a period of 24 weeks. They will also be invited to participate in sub-studies working on the analysis of gonioscopic images, detection of biomarkers for neovascular glaucoma and risk factors for ischaemic central retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria will be considered for enrolment to the trial:

* Male or female ≥ 18 years
* IOP in the study eye ≤ 21mmHg
* Primary ischaemic CRVO or conversion to ischaemic CRVO in the study eye for no longer than 4 weeks
* Best-corrected visual acuity (BCVA) ETDRS letter score < 35 (< 20/200 Snellen equivalent) in the study eye
* ≥ 10-disc area of retinal capillary obliteration on fluorescein fundus angiography in the study eye (central fundus: macular area as defined by the optic disc and the arcades, an approximate 6000 micron circle around the fovea) and/or large, confluent retinal haemorrhages in the study eye

Must be accompanied by 4 or more out of 6 following criteria:

* A relative afferent pupillary defect (with a normal fellow eye)
* ≥ 10 cotton-wool-spots in the study eye
* Venous tortuosity in the study eye
* Peripheral visual field defects corresponding to ischaemia (Goldmann perimeter or other semi-automatic kinetic methods) in the study eye
* Engorged vessels on iris and/or in the chamber angle in the study eye
* Detectable anterior chamber flare in the study eye

Exclusion Criteria:

Subjects presenting 1 or more of the following criteria will not be enrolled in the trial:

* Ocular conditions with a poorer prognosis in the fellow eye than in the study eye
* Primary or secondary glaucoma in the study eye
* Prior or concomitant ocular treatment with anti-VEGF in the study eye (ranibizumab/bevacizumab is not allowed within the last 45 days, aflibercept within the last 90 days) before screening visit
* Use of anti-VEGF treatment in the fellow eye during the trial
* Previous use of intraocular corticosteroids at any time or use of periocular corticosteroids in the study eye within 90 days prior to screening visit
* History of idiopathic or autoimmune uveitis in either eye
* Presence of NVD, NVE or anterior segment neovascularisation (NVA or NVI) in the study eye
* Previous PRP in the study eye
* Intraocular surgery (other than intravitreal anti-VEGF treatment) or laser treatment in the study eye within the past 90 days before screening visit
* Patients with a history of breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
NVG component | Week 24
  Co-primary I: NVG component scored dichotomously (NVG=yes/NVG=no) where "yes" is development of NVI, NVA, NVD, and/or NVE, or rescue treatment; "no" otherwise
IOP component | Week 24
  Co-primary II: IOP component scored dichotomously (failure/success); "failure" is rise in IOP from baseline to week 24 of ≥ 20% to > 21 or rescue treatment; "success" otherwise

SECONDARY OUTCOMES:
Secondary NVG | 24 weeks
  The time to development of secondary NVG in the study eye up to week 24 (in case aganirsen does not totally inhibit but slows down the development of NVG).
Anterior segment neovascularisation | 24 weeks
  The time to development of anterior segment neovascularisation (NVI or NVA), NVD or NVE in the study eye, requiring PRP or cryotherapy up to week 24.
NVG Classification | 24 weeks
  NVG Classification at 24 weeks on a scale from 1 (non-NVG) to 6 (most advanced NVG) based on central reading of neovascularisation
Visual Acuity | 24 weeks
  The change from baseline in BCVA (EDTRS letter score) in the study eye to week 24.
Number of additional needed laser treatments and re-treatments in the study eye at up to week 24 | 24 weeks
  Number of additional needed laser treatments and re-treatments in the study eye at up to week 24
Required intensity of laser spots of additional laser treatments and re-treatments in the study eye at up to week 24 | 24 weeks
  Required intensity of laser spots of additional laser treatments and re-treatments in the study eye at up to week 24
Retinal non-perfusion area | 24 weeks
  The change from baseline in size of retinal non-perfusion areas in the study eye to week 24
Retinal Thickness | 24 weeks
  Absolute change from baseline in retinal thickness in the study eye, assessed by spectral domain optical coherence tomography (SD-OCT) at week 24
Quality of Life | 24 weeks
  The change from baseline in the NEI-VFQ-25 health questionnaire total score to week 24
Quality of Life on EQ-5D | 24 weeks
  The change from baseline in the EQ-5D health questionnaire score to week 24
Safety: Incidence of treatment-emergent Adverse Events | 24 weeks
  Incidence, causality and intensity of adverse events between the treatment arms

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lorenz K, Scheller Y, Bell K, Grus F, Ponto KA, Bock F, Cursiefen C, Flach J, Gehring M, Peto T, Silva R, Tal Y, Pfeiffer N. A prospective, randomised, placebo-controlled, double-masked, three-armed, multicentre phase II/III trial for the Study of a Topical Treatment of Ischaemic Central Retinal Vein Occlusion to Prevent Neovascular Glaucoma - the STRONG study: study protocol for a randomised controlled trial. Trials. 2017 Mar 16;18(1):128. doi: 10.1186/s13063-017-1861-3. PMID 28302155